CLINICAL TRIAL: NCT05461495
Title: NYUCI-ES: Psychosocial Intervention to Improve Health Outcomes for Chinese and Korean ADRD Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: NYU Langone Health (Other); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P50MD017356-8241; P50MD017356 (NIH)
Record Dates: First submitted 2022-05-18; First posted 2022-07-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Dementia Caregivers; Diabetes; Heart Disease; Overweight
Keywords: Dementia caregivers; Social support; depressive symptoms; physical health; Chinese American; Korean American
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Overweight; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Treatment group will receive 6 counseling sessions, participate in local support group and on-line chat group, and receive "ad hoc" counseling.
  Interventions: Behavioral: Treatment Group
- Control Group (No Intervention): Control group will participate in on-line chat group, and call the counselor for resource information and support as needed.

INTERVENTIONS:
Behavioral: Treatment Group — This intervention is unique in its emphasis on family support and in providing ongoing availability of the counselor. While the NYUCI is being implemented in several communities, its effectiveness in Chinese and Korean American dementia caregivers has not been tested. The first component of the intervention consists of two individual and four family counseling sessions that include relatives suggested by the caregiver. The second component of the intervention is participation in a support group to provide the caregiver with continuous emotional support and education. The third component of the treatment is participation in an on-line chat group to provide peer support. The fourth component of the treatment is "ad hoc" counseling the continuous availability of counselors to caregivers and families to help them deal with crises and with the changing nature and severity of their relatives' symptoms over the course of the disease.
  Arms: Treatment Group

SUMMARY:
This study will conduct a two-arm randomized controlled trial to test the efficacy of a culturally tailored version of the NYU Caregiver Intervention (NYUCI) plus enhanced support (ES) through online chat groups (the NYUCI plus WeChat/Kakaotalk/other social media apps [popular social media apps for individuals of Chinese or Korean descents] peer support which we call the NYUCI-ES in reducing health risks for cardiometabolic disease among older Chinese and Korean American adults caring for relatives with ADRD. In collaboration with community organizations across the New York and northern New Jersey metropolitan area, we will enroll 300 caregivers of people with ADRD (150 Chinese and 150 Korean) in this study. Aim 1: Develop culturally adapted informational and educational materials about dementia and caregiving issues for social service providers of the intervention and for family caregivers. Aim 2: Test the hypothesis, H1: A counseling and support intervention (the NYUCI-ES) will significantly improve psychosocial factors such as depression, stress self-rated health and chronic disease management among Chinese and Korean-American ADRD caregivers and these changes will be mediated by improvement in social support. H1a: By the first (6- month) follow-up, the mediators (increases in social support, stress reaction) will improve significantly in the intervention group compared to baseline values and the control group. H1b: These improvements will be maintained, and lead to reduction in depressive symptoms, and improvement in self-reported health and chronic disease self-management by the 12-month follow-up compared to the control group. Aim 3: Test the hypothesis, H2: the NYUCI-ES will reduce biologic risk factors, including metabolic health (glycosylated hemoglobin, BMI) and inflammation (hsCRP, lipid metabolism, etc.) within 6 months of enrollment compared to baseline and a control group; these changes will be mediated through increases in social support and decreases in depressive symptoms and will be maintained at the 12-month follow-up. The public health significance of these findings will likely have an impact on health care policy for CGs from diverse underserved ethnic and cultural backgrounds, potentially reducing morbidity, and improving their quality of life.

DETAILED DESCRIPTION:
The physical and emotional demands of dementia caregiving can have enormous negative effects on caregivers' physical and mental health. Dementia caregivers have increased risk of hypertension and diabetes, compared to non-caregivers, especially in minority populations. The NYUCI has proven efficacy in reducing psychological outcomes among largely White samples of caregivers of persons with ADRD and has been widely replicated and translated in the USA and elsewhere. This study will provide the first large- scale test of the potential effects of the NYUCI-ES, a multicomponent intervention that includes individual and family counseling and ongoing support via support group and online chat groups and ad hoc (on demand) counseling.

Chinese American and Korean American dementia caregivers with multiple chronic conditions will be enrolled. This is an unblinded, randomized trial to assess the effectiveness of NYUCI intervention among Chinese and Korean American dementia caregivers. The study will utilize quantitative methods to learn more about the physical health and psychological health outcomes in Chinese and Korean American dementia caregivers.

This study lasts 1 year. The intervention will include two group with each ethnicity group. All participants will participate an on-line chat group and call the counselor for resource information and support as needed. Participants in the treatment group will receive 6 counseling sessions an participate in local support group.

ELIGIBILITY:
Inclusion Criteria:

* A spouse or other family caregiver of Chinese or Korean ancestry living in New York City or Bergen County New Jersey, who is willing to participate in the study (additional family members can be included in family counseling sessions if the CG is assigned to the treatment group)
* at least 50 years of age
* self-identified as a primary caregiver
* have access to Internet and phone with SMS and voice messaging
* no plans to move for 12 months
* able to read English, Chinese, or Korean
* capable of completing informed consent
* meet specific cardiometabolic and depressive symptom criteria: Cardiometabolic syndrome: It will not be required to submit objective measurement of cardiometabolic disorder, self-reported medical conditions will be accepted for enrollment. Diabetes: self-reported OR A1C >= 5.7% OR High Cholesterol: self-reported OR low-density lipoprotein (LDL) > 130 mg/dL or total cholesterol > 200 mg/dL (American Heart Association 2018) OR Hypertension: self-reported OR systolic blood pressure (SBP) >= 130 mmHg or diastolic blood pressure (DBP) >= 80mmHg (2017 ACC/AHA hypertension guideline) OR Body Mass Index > 23 kg/m2 by self-reported or measured height and weight (WHO expert consultation regarding Asian cut-off) OR other related metabolic syndrome, such as euthyroid hypothyroxinemia
* care recipient regularly has trouble remembering recent events, repeat the same question over and over, or lose or misplace things

Exclusion Criteria:

* current alcoholic or substance abuse; and history of psychiatric diagnoses requiring hospitalization during the past 5 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 12 months
  Depressive symptoms will be assessed using the 9-item Patient Health Questionnaire-9 (PHQ-9),because of its brevity, well-validated reliable measures, that has been used in other studies of Chinese and Korean adults.
Self-rated Health | 12 months
  This measure includes three global self-rated physical health items from the Older Americans Resources and Services (OARS) battery of questionnaires (ICC = 0.83) to assess subjective evaluation of health. The sum of the 3 questions is used to measure self-rated health.
Caregiving related stress | 12 months
  It will be measured by the severity of reaction axis of the Revised Memory and Behavior Problems Checklist.
Chronic disease self management behaviors | 12 months
  It will be measured with the Summary of Diabetes Self-Care Activities Measure, which is widely used by diabetes researchers and assesses frequency of healthy eating (e.g., how many of the last seven days did you eat five or more servings of fruits and vegetables), exercise, testing blood sugar, foot care, and smoking.
Social support | 12 months
  The following measures will be used to assess various aspects of social support. Subjective social support will be measured using the Lubben Social Network Scale-6-item version. The Social Support Availability Scale will be used to evaluate the availability of emotional, instrumental, and informational support. The use of formal support services, such as respite care, support groups, and home health care aids, will be assessed with the Service Utilization Scale. Additionally, the WeChat Use Intensity Questionnaire (WUIQ) will be used to measure the use of social media applications, and it will be adapted to include KakaoTalk and other platforms.
Diabetes | 12 months
  HbA1C will be measured through a fingerstick and processed in the Bayer A1CNow® device, which is National Glycohemoglobin Standardization Program Certified and has demonstrated accuracy and precision. A cut-off of HbA1C >= 5.7% will be used to determine pre-diabetic status.
Lipid metabolism | 12 months
  Triglycerides, Cholesterol, HDL, LDL, and VLDL will be measured along with HbA1c using the same method. Low-density lipoprotein (LDL) > 130 mg/dL or total cholesterol > 200 mg/dL will be used to determine high cholesterol.
Hypertension | 12 months
  Blood pressure will be measured utilizing PhenX Toolkit recommended procedures and OMRON automated blood pressure machine. A cut-off of systolic blood pressure (SBP) >= 130 mmHg or diastolic blood pressure (DBP) >= 80mmHg will be used to determine the presence of hypertension
Waist circumferences and Body Mass index (BMI) | 12 months
  Waist circumference will be measured using a flexible, non-stretchable measuring tape at the halfway point between the lower margin of the last palpable rib and the top of the hip bone. BMI will be measured through height (feet/inches or cm) and weight (lb or kg) measurements. A digital scale and stadiometer will be used to measure height and weight. Weight and height will be combined to report Body Mass Index in > 23 kg/m2 will be used to determine obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Bei Wu, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data collected during the trial will be shared between 9 months and 36 months following article publication or as required by a condition of awards and agreements supporting the research, for researchers who provide a methodologically sound proposal. Data will be made available at https://www.icpsr.umich.edu/web/pages (Note: a specific link will be provided after the study is published/when the DOI is obtained.) The protocol, statistical analysis plan, and analytic code will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Data will be made available at Clinicaltrials.gov and ICPSR (a specific link will be provided after the study is published/when the DOI is obtained).

REFERENCES:
- [Background] Wang J, Leong IT, Johnson MK, Pei Y, Lee KH, Mittelman MS, Epstein C, Cho S, Wu B. What Matters to Chinese and Korean American Dementia Caregivers: Navigating Cultural Influences in Dementia Care from Caregivers' Perspectives. J Alzheimers Dis. 2024;98(2):519-538. doi: 10.3233/JAD-231140. PMID 38427483